CLINICAL TRIAL: NCT02337439
Title: Cognitive Remediation for Perceptual Deficits in Schizophrenia
Brief Title: Perceptual Deficits in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V1CDA2013-24; 01856 (Other: VACHS IRB)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensory Information Processing Training (Experimental): Computerized training designed to improve sensory processing
  Interventions: Behavioral: Sensory Information Processing Training
- Active Control Training (Active Comparator): Commercially available computer exercises that were not designed specifically to improve sensory information processing.
  Interventions: Behavioral: Active Control Training

INTERVENTIONS:
Behavioral: Sensory Information Processing Training — Computer exercises requiring identification of visual stimuli on computer screen and response with keyboard
  Arms: Sensory Information Processing Training
Behavioral: Active Control Training — Commercially available educational software
  Arms: Active Control Training

SUMMARY:
In this study, participants with schizophrenia and schizoaffective are given computer exercises to complete. The goals of the study are to determine whether: 1) any of the computer exercises can improve information processing problems in schizophrenia, 2) improvements in information processing are related to other cognitive improvements, and 3) there are changes in brain activity associated with using the computer exercises.

The study will involve clinical interviews, cognitive tests, and frequent computerized cognitive training over the course of 2 months. Some participants will also have electroencephalography, a non-invasive test that measures brain activity, to determine whether there are changes in brain activity with the computer training.

DETAILED DESCRIPTION:
Schizophrenia is a disabling neurodevelopmental illness, affecting nearly 1% of the population. The disability of schizophrenia is due in large part to the effects of the illness on cognitive faculties. Current medications for schizophrenia do not generally improve cognition, so a major contribution to disability remains undertreated. Computerized cognitive remediation programs, which produce activity-dependent recruitment of neural resources to specifically enhance under-functioning brain systems, have been effective at improving both cognition and community functioning in patients with schizophrenia, but the effects are still modest. Our preliminary work has suggested that our training is associated with improvements in visual memory, though visual memory has been a cognitive area more refractory to cognitive training.

In this study, participants with schizophrenia or schizoaffective disorder will be randomized to receive different computer exercises to help determine whether computer exercises can improve memory in schizophrenia, and whether the cognitive training is associated with changes in neural activity.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or schizoaffective disorder
* English speaking and reading

Exclusion Criteria:

* current substance abuse
* visual impairment
* neurological conditions
* current enrollment in another research study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive test performance | up to 6 months
  Neuropsychological testing

SECONDARY OUTCOMES:
Psychiatric symptoms | up to 6 months
  Clinical interviews and ratings
Social Functioning | up to 6 months
  Clinical rating scales

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Tandon R, Keshavan MS, Nasrallah HA. Schizophrenia, "just the facts" what we know in 2008. 2. Epidemiology and etiology. Schizophr Res. 2008 Jul;102(1-3):1-18. doi: 10.1016/j.schres.2008.04.011. Epub 2008 Jun 2. PMID 18514488
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Carpenter WT, Buchanan RW. Lessons to take home from CATIE. Psychiatr Serv. 2008 May;59(5):523-5. doi: 10.1176/ps.2008.59.5.523. PMID 18451009
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461
- [Background] Surti TS, Wexler BE. A pilot and feasibility study of computer-based training for visual processing deficits in schizophrenia. Schizophr Res. 2012 Dec;142(1-3):248-9. doi: 10.1016/j.schres.2012.09.013. Epub 2012 Oct 6. No abstract available. PMID 23043873